CLINICAL TRIAL: NCT00334919
Title: Randomized Clinical Trial of the Naturopathic Anti-Inflammatory Diet
Brief Title: RCT of the Naturopathic Anti-Inflammatory Diet
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Patricia Elmer, PhD, Helfgott Research Institute
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21AT002374-01A1 (NIH); R21AT002374-01A1 (NIH)
Record Dates: First submitted 2006-06-06; First posted 2006-06-08 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2009-05

CONDITIONS: Diabetes Mellitus, Type 2; Prediabetes
Keywords: Diabetes; Pre-Diabetes; Anti-Inflammatory Diet; Diet Study; Inflammation; Diabetic Diet
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Diabetes Mellitus; Glucose Intolerance; Inflammation | interventions — Diet; Anti-Inflammatory Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Diet (Anti-Inflammatory or standard diabetic diet) — 6 weeks standard ADA diet, then randomized to either ADA or antiinflammatory (AI) diet for 6 weeks

SUMMARY:
The purpose of this study is to determine if the naturopathic Anti-Inflammatory Diet results in reduced inflammation and a better response by the immune system when compared to a standard diabetic diet based on the current American Diabetes Association guidelines.

DETAILED DESCRIPTION:
This study will test the effects of two different diets on the immune system and inflammation in diabetes and pre-diabetes. These diets are the "Anti-Inflammatory Diet" (AI Diet) used by many naturopathic doctors and a standard diabetic diet based on the American Diabetes Association recommendations (ADA Diet). The AI diet excludes wheat, dairy products, eggs, red meat, caffeine, alcohol, peanuts and certain fruits and vegetables. The ADA diet includes most foods but controls the amount of each of the food groups.

Naturopathic physicians often use healthful diets to treat diseases but many of these diets have not been compared to usual medical diet treatments. We will be looking at blood markers that show how the immune system responds to the different diets. We are expecting that the AI diet will result in less inflammation and a better response by the immune system than the ADA diet. We will also be looking at levels of blood lipids and glucose to see any effects on these risk factors.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 25-45 kg/m2
* Age 18-75 yrs
* Diagnosed with type 2 diabetes or pre-diabetes
* At risk for type 2 diabetes. Must meet 2 of the following 3 criteria: BMI 30-45 kg/m2, age 50 or older, and/or family history of type 2 diabetes
* Fasting blood glucose of 100-200 mg/dl
* Provide informed consent

Exclusion Criteria:

* Current major debilitating mental or physical illness that would interfere with participation (as determined by the participant's medical history)
* Taking diabetic medication other than sulfonylurea
* Taking Gymnema silvestra (a naturopathic diabetes treatment)
* Taking medications that have anti-inflammatory affects (lipid lowering agents, NSAIDS, COX 2 inhibitors, aspirin, HRT, oral contraceptives, testosterone, seizure medications)
* Taking weight loss medications
* Severe renal, hepatic, or heart disease
* Triglycerides >500 mg/dL
* Bulimia
* Pregnancy or lactation
* Current excessive use of alcohol
* Current/recent chronic use of recreational drugs
* Smoker
* More than 4 hours/week of aerobic exercise
* Have gained or lost more than 15 pounds during previous 6 months
* Planning on moving out of the area in the next 4 months
* Is a participant in another medical research study
* Is following a weight loss diet
* Is unwilling to accept random assignment of the experimental diets
* Food preferences and/or allergies that will interfere with consumption of experimental diet

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Cytokines | 13 weeks

SECONDARY OUTCOMES:
Glucose | 113 weeks
Weight | 13 weeks
Lipids | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Elmer, PhD, Principal Investigator — National College of Naturopathic Medicine
Locations (1):
- Oregon Health & Science University General Clinical Research Center, Portland, Oregon, United States